CLINICAL TRIAL: NCT04348175
Title: A Phase 1, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics of Setmelanotide in Subjects With Varying Degrees of Renal Impairment
Brief Title: A Phase 1 Study to Evaluate the Pharmacokinetics of Setmelanotide in Subjects With Varying Degrees of Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: RM-493-029
Record Dates: First submitted 2020-03-30; First posted 2020-04-16 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — setmelanotide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Mild impairment (Experimental)
  Interventions: Drug: Setmelanotide
- Moderate impairment (Experimental)
  Interventions: Drug: Setmelanotide
- Severe impairment (Experimental)
  Interventions: Drug: Setmelanotide
- Normal (control) (Experimental)
  Interventions: Drug: Setmelanotide

INTERVENTIONS:
Drug: Setmelanotide — Setmelanotide will be administered as a single SC dose of 2.0 mg on Day 1. A dose higher than 2.0 mg will not be used during the study. Dose may be lowered based on safety data.

SUMMARY:
This is a Phase 1, multi-center, open-label, single-dose study designed to assess the effect of renal impairment on the PK of setmelanotide. A total of approximately 32 subjects (approximately 8 subjects in each renal impairment group and 8 healthy subjects with normal renal function) are planned to be enrolled across 4 centers in the United States. At screening, subjects will be assigned to a study group according to eGFR.

Cohort A - Mild Renal Impairment

Cohort B - Moderate Renal Impairment

Cohort C - Severe Renal Impairment

Cohort D - Normal Renal Function (control)

ELIGIBILITY:
Inclusion Criteria:

1. The subject is male or female 18 to 83 years of age, inclusive.
2. The subject has a BMI of 22 to 40 kg/m2, inclusive, at screening.
3. Female subjects of childbearing potential must use an acceptable method of birth control (ie, diaphragm with spermicide, intrauterine device, condom with foam or vaginal spermicide, oral contraceptives, or abstinence) or be surgically sterile (ie, hysterectomy, bilateral tubal ligation or bilateral oophorectomy), or postmenopausal (defined as amenorrhea 12 consecutive months and documented plasma follicle-stimulating hormone level in the postmenopausal range according to the laboratory used). Female subjects must have a negative pregnancy test at screening and before the first dose of study drug and must not be lactating.

   Male subjects with female partners of childbearing potential must be vasectomized, be willing to use an acceptable method of birth control, or practice abstinence during the study. Male subjects must not donate sperm during and for 90 days following their participation in the study.
4. The subject agrees to comply with all protocol requirements.
5. The subject is able to provide written informed consent.

   Additional Inclusion Criteria for Subjects with Renal Impairment Only (Cohorts A, B, and C):
6. The subject has mild, moderate, or severe renal impairment as determined by eGFR and calculated using the MDRD formula.
7. The subject's renal insufficiency or other related concomitant medical conditions (eg, hypertension, diabetes, anemia) have remained stable for at least 3 months before study drug dosing.
8. The subject has a resting blood pressure of 90 to 165 mm Hg (systolic) and 45 to 100 mm Hg (diastolic). Measurement can be repeated if the subject has an elevated value that is not consistent with previous history.
9. The subject has a QTcF of <500 msec.
10. The subject is judged by the investigator to be in good general health, as determined by medical history, clinical laboratory assessments, vital sign measurements, 12-lead ECG results, and physical examination findings, except for findings that, as judged by the investigator, are consistent with the subject's renal impairment or other stable concomitant medical conditions.

    Additional Inclusion Criteria for Healthy Subjects Only (Cohort D):
11. The subject has normal renal function (≥90 mL/min) as determined by eGFR calculated using the MDRD formula.
12. The subject will be "matched" to previous Cohorts A, B, and C with regards to age, sex, and BMI characteristics. Each subject in Cohort D will be within 20% of the median age and BMI of the combined median age and BMI across Cohorts A, B, and C.
13. The subject has a resting blood pressure of 90 to 150 mm Hg (systolic) and 40 to 100 mm Hg (diastolic).
14. The subject is judged by the investigator to be in good general health, as determined by medical history, clinical laboratory assessments, vital sign measurements, 12-lead ECG results, and physical examination findings.

Exclusion Criteria:

1. The subject has a history or clinical manifestations of a significant neurological, cardiovascular, gastrointestinal, pulmonary, hematologic, immunologic, hepatic, genitourinary, endocrine, metabolic, or psychiatric disease that would preclude study participation, as judged by the investigator.
2. The subject has a positive test result for human immunodeficiency virus Types 1 or 2 antibodies or hepatitis B surface antigen at screening.
3. The subject has a history of alcoholism or drug abuse within 3 months before screening.
4. The subject is unable or unwilling to abstain from alcohol, marijuana and related substances, caffeine, cigarette smoking, vaping, or any form of tobacco or nicotine from 48 hours prior to study drug dosing until completing study assessments on Day 5.
5. The subject is involved in strenuous activity or contact sports within 24 hours of the first dose of study drug or during the study.
6. The subject has donated blood or blood products >450 mL within 30 days before the first dose of study drug.
7. The subject has a history of relevant drug and/or food allergies (ie, allergy to setmelanotide or any excipients, or any significant food allergy).
8. The subject has used prescription drugs from 1 week prior to randomization and throughout the study, except for prescription medications used for the treatment of stable concomitant conditions; examples include the following: diabetes, hypertension, hypercholesterolemia, hyperlipidemia or hypothyroidism. Medications used to treat these indications are allowed, so long as the subject has been on a stable dose for at least 2 weeks prior to randomization and plans to continue a stable dose throughout the study.
9. The subject has received study drug in another investigational study within 30 days of dosing.
10. The subject has a positive test result for drugs of abuse (including marijuana, and except positive test results associated with prescription medications that have been reviewed and approved by the investigator) or alcohol at screening or before the first dose of study drug.
11. The subject has ALT or AST >2 × ULN at screening.
12. The subject has HbA1c >10%. With Sponsor approval, a subject who has a HbA1c >10% may be enrolled into the study if, in the opinion of the primary investigator, the subject's diabetes is reasonably controlled and the subject is otherwise appropriate for this study.
13. The subject has any personal history of cancer (unless stable and in remission for ≥5 years), multiple atypical nevi, nevoid basal cell carcinoma syndrome, or nonmelanoma skin cancer requiring treatment beyond local excision.
14. The subject has any close family history (parents or siblings) of melanoma.
15. The subject has significant dermatologic findings relating to melanoma or premelanoma skin lesions, determined as part of a screening comprehensive skin evaluation performed by a qualified dermatologist, the principle investigator, or a nurse practitioner (ordered by preference) . Any concerning lesions identified during screening will be biopsied and results known to be benign prior to enrollment. If the pretreatment biopsy results are of concern, the subject may need to be excluded from the study.
16. The subject has history of clinically significant recent surgery (within 60 days of screening).
17. The subject has current or recent (within last month) infection or viral illness.
18. In the opinion of the investigator, the subject is not suitable for entry into the study.

    Additional Exclusion Criteria for Subjects with Renal Impairment Only (Cohorts A, B, and C):
19. The subject has a positive test result for antibodies to hepatitis C virus with evidence of viral load at screening.
20. The subject has nephrotic syndrome, defined as urine dipstick 4+ for protein and plasma albumin <3.0 g/dL, and then confirmed if proteinuria >5 g/day.
21. The subject has renal impairment due to rapidly growing, space-occupying lesions (eg, carcinoma of the kidney, tuberculosis).
22. Subject has a history of renal transplant.
23. The subject has a hemoglobin value less than 8.0 g/dL.
24. The subject has a clinically relevant immunologic disease.

    Additional Exclusion Criteria for Healthy Subjects Only (Cohort D):
25. The subject has a positive test result for antibodies to hepatitis C virus at screening.

Ages: 18 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2021-04-17 (Actual); Study Completion 2021-04-17 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Parameter - Peak Plasma Concentration (Cmax) | 5 days
  The primary objective of this study is to evaluate the PK of a single dose of Setmelanotide administered SC in subjects with varying degrees of renal impairment and that of healthy matched control subjects.
Pharmacokinetic Parameter - Area under the plasma concentration versus time curve (AUC) | 5 days
  The primary objective of this study is to evaluate the PK of a single dose of Setmelanotide administered SC in subjects with varying degrees of renal impairment and that of healthy matched control subjects.

SECONDARY OUTCOMES:
Number of Participants with Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | 5 days
  The secondary objective of this study is to evaluate the safety and tolerability of a single dose of Setmelanotide administered SC in subjects with varying degrees of renal impairment.
Number of Participants with Abnormal Vital Sign Findings | 5 days
  Vital signs will include systolic and diastolic blood pressure, pulse rate, respiratory rate, and body temperature.
Number of subjects with Abnormal Electrocardiogram (ECG) findings | 5 days
  Electrocardiogram assessments will include comments on whether the tracings are normal or abnormal, rhythm, presence of arrhythmia or conduction defects, wave morphology, any evidence of myocardial infarction, or ST-segment, T-Wave, and U Wave abnormalities.
Number of subjects with Abnormal Findings in Physical Examination | 5 days
  A full physical examination will include, at minimum, assessment of skin, head, ears, eyes, nose, throat, neck, thyroid, lungs, heart, cardiovascular, abdomen, lymph nodes, and musculoskeletal system/extremities.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Marshfield Clinic Research Institute, Marshfield, Wisconsin